CLINICAL TRIAL: NCT05646862
Title: A Phase III, Multicenter, Randomized, Open-Label Study Evaluating the Efficacy and Safety of Inavolisib Plus Fulvestrant Versus Alpelisib Plus Fulvestrant in Patients With Hormone Receptor-Positive, HER2-Negative, PIK3CA Mutated, Locally Advanced or Metastatic Breast Cancer Who Progressed During or After CDK4/6 Inhibitor and Endocrine Combination Therapy
Brief Title: A Study Evaluating the Efficacy and Safety of Inavolisib Plus Fulvestrant Compared With Alpelisib Plus Fulvestrant in Participants With HR-Positive, HER2-Negative, PIK3CA Mutated, Locally Advanced or Metastatic Breast Cancer Post CDK4/6i and Endocrine Combination Therapy
Acronym: INAVO121
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO43919; 2022-502322-41-00 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib; Fulvestrant; Alpelisib; Bupropion; Omeprazole; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inavolisib + Fulvestrant (Experimental): Participants will be administered the treatments as outlined in the interventions section.
  Interventions: Drug: Inavolisib; Drug: Fulvestrant
- Alpelisib + Fulvestrant (Active Comparator): Participants will be administered the treatments as outlined in the interventions section.
  Interventions: Drug: Fulvestrant; Drug: Alpelisib
- Sub-study: Inavolisib + Fulvestrant + CYP substrates (Experimental): Participants will be administered the treatments as outlined in the interventions section.
  Interventions: Drug: Inavolisib; Drug: Fulvestrant; Drug: Bupropion; Drug: Omeprazole; Drug: Midazolam

INTERVENTIONS:
Drug: Inavolisib — Participants will be administered a 9 milligram (mg) inavolisib tablet orally once a day (PO QD) on Days 1-28 of each 28-day cycle of main study and sub-study.
  Arms: Inavolisib + Fulvestrant; Sub-study: Inavolisib + Fulvestrant + CYP substrates
Drug: Fulvestrant — Participants will be administered 500 mg of fulvestrant on Days 1 and 15 of Cycle 1 and then on Day 1 of each subsequent 28-day cycle of main study and sub-study.
Drug: Alpelisib — Alpelisib will be administered to participants at the approved dose in combination with fulvestrant: 300 mg taken PO QD and on days 1-28 of each 28-day cycle.
  Arms: Alpelisib + Fulvestrant
Drug: Bupropion — Participants will be administered bupropion PO on Day -3 and Day 12 of Cycle 1 of the sub-study.
  Arms: Sub-study: Inavolisib + Fulvestrant + CYP substrates
Drug: Omeprazole — Participants will be administered omerprazole PO on Day -4 and Day 11 of Cycle 1 of sub-study.
  Arms: Sub-study: Inavolisib + Fulvestrant + CYP substrates
Drug: Midazolam — Participants will be administered midazolam PO on Day -4 and Day 11 of Cycle 1 of sub-study.
  Arms: Sub-study: Inavolisib + Fulvestrant + CYP substrates

SUMMARY:
This is a Phase III, multicenter, randomized, open-label, global study designed to evaluate the efficacy and safety of inavolisib plus fulvestrant compared with alpelisib plus fulvestrant in patients with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2) -negative, PIK3CA-mutated, locally advanced (LA) or metastatic breast cancer (mBC), who progressed during or after cyclin dependent kinase 4/6i (CDK4/6i)-based therapy.

DETAILED DESCRIPTION:
The drug-drug interaction (DDI) substudy will evaluate the impact of repeat doses of inavolisib (coadministered with fulvestrant) on single-dose pharmacokinetics of sensitive CYP450 enzyme substrates (midazolam, omeprazole and bupropion) in participants with hormone receptor (HR)-positive, HER2-negative, PIK3CA-mutated, locally advanced (LA) or metastatic breast cancer (mBC), who progressed during or after CDK4/6 inhibitor (CDK4/6i) in combination with endocrine therapy (ET).

ELIGIBILITY:
Inclusion Criteria for Main Study and Sub-study:

* If pre/perimenopausal women and men treatment with luteinizing hormone-releasing hormone (LHRH) agonist therapy beginning at least 2 weeks prior to Day 1 of Cycle 1
* Histologically or cytologically confirmed adenocarcinoma of the breast that is locally advanced or metastatic and is not amenable to surgical or radiation therapy with curative intent
* Documented HR +/ HER2- tumor according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines
* Confirmation of biomarker eligibility: detection of specified mutation(s) of PIK3CA via specified test
* Disease progression after or during treatment with a combination of CDK4/6i and endocrine therapy: <= 2 prior lines of systemic therapy in mBC setting; CDK4/6i based therapy does not need to be the last one received prior study entry; one line of chemotherapy in mBC setting allowed
* Measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Participants for whom endocrine-based therapy is recommended and treatment with cytotoxic chemotherapy is not indicated at time of entry into the study, as per national or local treatment guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Life expectancy of > 6 months
* Adequate hematologic and organ function prior to initiation of study treatment

Exclusion Criteria for both Main Study and Sub-study:

* Metaplastic breast cancer
* Prior treatment in locally advanced or metastatic setting with any PI3K, AKT, or mTOR inhibitor or any agent whose mechanism of action is to inhibit the PI3K/-AKT/-mTOR pathway
* Participant who relapsed with documented evidence of progression > 12 months from completion of adjuvant CDK4/6i based therapy with no treatment for metastatic disease
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes
* Inability or unwillingness to swallow pills
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Any history of leptomeningeal disease or carcinomatous meningitis
* Known and untreated, or active central nervous system (CNS) metastases. Participants with a history of treated CNS metastases are eligible if they meet specific certain criteria
* Any concurrent ocular or intraocular condition that, in the opinion of the investigator, would require medical or surgical intervention during the study period to prevent or treat vision loss that might result from that condition
* Active inflammatory or infectious conditions in either eye or history of idiopathic or autoimmune-associated uveitis in either eye
* Requirement for daily supplemental oxygen
* Symptomatic active lung disease, including pneumonitis
* History of or active inflammatory bowel disease
* Any active bowel inflammation
* Clinically significant and active liver disease, including severe liver impairment, viral or other hepatitis, current alcohol abuse, or cirrhosis
* Participants with known human immunodeficiency virus infection that meet specific criteria
* History of other malignancy within 5 years prior to screening, except for cancers with very low risk of recurrence
* Chronic therapy of >= 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressants for a chronic disease
* Active ongoing osteonecrosis of the jaw

Exclusion Criteria for Main Study Only:

* Pregnant, lactating, or breastfeeding, or intending to become pregnant during the study or at least 60 days after the final dose of study treatment
* Known active, systemic infection at study enrollment, or any major episode of infection requiring treatment with intravenous antibiotics or hospitalization within 7 days prior to Day 1 of Cycle 1
* Investigational drug(s) within 4 weeks before randomization or within 5 half-lives of the investigational drug(s), whichever is longer
* Allergy or hypersensitivity to components or excipients of the inavolisib, fulvestrant, or alpelisib formulations
* History of severe cutaneous reactions like Stevens-Johnson Syndrome, Erythema Multiforme, Toxic Epidermal Necrolysis, or Drug Reaction with Eosinphilia and Systemic Symptoms

Exclusion Criteria for Sub-study Only:

* Pregnant, lactating, or breastfeeding, or intending to become pregnant during the substudy or within 2 weeks after the final dose of inavolisib and within 2 years after the final dose of fulvestrant, whichever is longer
* Known active, systemic infection at study enrollment, or any major episode of infection requiring treatment with intravenous antibiotics or hospitalization within 7 days prior to Day -4 of Cycle 1
* Investigational drug(s) within 4 weeks prior to Day -4 or within 5 half-lives of the investigational drug(s), whichever is longer
* Allergy or hypersensitivity to components or excipients of the inavolisib, fulvestrant formulations
* Treatment with mild, moderate, or strong inducers of CYP2B6, CYP3A4, and/or CYP2C19 (including St. John's Wort) within 14 days or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study treatment on Day -4 until after the final PK sample has been collected on Day 15 of Cycle 1
* Treatment with mild, moderate, or strong inhibitors of CYP2B6, CYP3A4, and/or CYP2C19 (including grapefruit juice or supplements) within 14 days or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study treatment on Day -4 until after the final PK sample has been collected on Day 15 of Cycle 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Blinded Independent Central Review (BICR)-Assessed Progression Free Survival (PFS) | From randomization until disease progression or death due to any cause (up to approximately 64 months)
Sub-study: Maximum observed Drug Concentration (Cmax) for Midazolam | Day -4 and -3 of Cycle (C) 1, Day (D) 11 and C1D12. A cycle is 28 days.
Sub-study: Cmax for Bupropion | Day -3, -2, -1 of C1D1, C1D12, C1D13, C1D14 and C1D15. A cycle is 28 days.
Sub-study: Cmax for Omeprazole | Day -4 and -3 of C1D11 and C1D12. A cycle is 28 days.
Sub-study: Area Under the Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUC [0-last]) for Midazolam | Day -4 and -3 of C1D11 and C1D12. A cycle is 28 days.
Sub-study: AUC (0-last) for Bupropion | Day -3, -2, -1 of C1D1, C1D12, C1D13, C1D14 and C1D15. A cycle is 28 days.
Sub-study: AUC (0-last) for Omeprazole | Day -4 and -3 of C1D11 and C1D12. A cycle is 28 days.
Sub-study: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC [0-infinity]) for Midazolam | Day -4 and -3 of C1D11 and C1D12. A cycle is 28 days.
Sub-study: AUC (0-infinity) for Bupropion | Day -3, -2, -1 of C1D1, C1D12, C1D13, C1D14 and C1D15. A cycle is 28 days.
Sub-study: AUC (0-infinity) for Omeprazole | Day -4 and -3 of C1D11 and C1D12. A cycle is 28 days.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization until death due to any cause (up to approximately 85 months)
BICR-Assessed Overall Response Rate (ORR) | Up to approximately 64 months
BICR-Assessed Best Overall Response (BOR) | Up to approximately 64 months
BICR-Assessed Clinical Benefit Rate (CBR) | Up to approximately 64 months
BICR-Assessed Duration of Response (DOR) | From CR or PR until disease progression or death due to any cause (up to approximately 64 months)
Time to Confirmed Deterioration (TTCD) in Pain | Day 1 of Cycles 1 and 2 and beyond, 30-day safety follow up visit, post-treatment tumor assessment follow-up with PRO collection and survival follow up visit (up to approximately 85 months). Each cycle is 28 days.
TTCD in Physical Functioning | Day 1 of Cycles 1 and 2 and beyond, 30-day safety follow up visit, post-treatment tumor assessment follow-up with PRO collection and survival follow up visit (up to approximately 85 months). Each cycle is 28 days.
TTCD in Role Functioning | Day 1 of Cycles 1 and 2 and beyond, 30-day safety follow up visit, post-treatment tumor assessment follow-up with PRO collection and survival follow up visit (up to approximately 85 months). Each cycle is 28 days.
TTCD in Global Health Status/Quality of Life (QOL) | Day 1 of Cycles 1 and 2 and beyond, 30-day safety follow up visit, post-treatment tumor assessment follow-up with PRO collection and survival follow up visit (up to approximately 85 months). Each cycle is 28 days.
Percentage of Participants with Adverse Events | Day 1 until 30 days after the final dose of study treatment (up to approximately 85 months)
Plasma Concentration of Inavolisib at Specified Timepoints | Day 1 and 15 of Cycle 1, and Day 1 of Cycles 2 and 3. Each cycle is 28 days.
Sub-study: Percentage of Participants with Adverse Events | Day -4 until 30 days after the final dose of study treatment (up to approximately 85 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (145):
- United States (14):
  - Cancer Blood and Specialty Clinic, Los Alamitos, California
  - Los Angeles Cancer Network, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Cleveland Clinic Florida, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Midtown West Medical, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute at Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Minnesota Oncology Hematology, Saint Paul, Minnesota
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
- Argentina (7):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
  - Fundacion CORI para la Investigacion y Prevencion del Cancer, La Rioja
  - Instituto de Oncología de Rosario, Rosario
  - Hosp Provincial D. Centenarios, Rosario
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Clinica Viedma S.A., Viedma
- Australia (7):
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - Bendigo Cancer Centre, Bendigo, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Belgium (6):
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Les Viviers, Charleroi
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Clinique Ste-Elisabeth, Namur
- Brazil (8):
  - NUPEC, Belo Horizonte, Minas Gerais
  - Hospital Santa Cruz / Centro de Oncologia D'Or, Curitiba, Paraná
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Instituto D?Or de Pesquisa e Ensino ? Hospital Esperança Recife, Recife, Pernambuco
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
- Canada (10):
  - Arthur J.E. Child Comprehensive Cancer Center-Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer ? Vancouver, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Juravinski Hospital, Hamilton, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - CIUSSS de l Est de l Ile de Montreal - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec
- China (14):
  - The First Hospital of Jilin University, Changchun
  - Sichuan Provincial Cancer Hospital, Chengdu
  - Sun yat-sen University Cancer Center, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Harbin Medical University Tumor Hospital, Harbin
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Tianjin Cancer Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Zhejiang Cancer Hospital, Zhejiang
- France (5):
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Centre Leon Berard, Lyon
  - ICM, Montpellier
  - Centre Eugene Marquis, Rennes
  - IUCT Oncopole, Toulouse
- Germany (9):
  - Uniklinik RWTH Aachen Klinik für Gynäkologie und Geburtsmedizin, Aachen
  - Universitätsklinikum Essen, Essen
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - Medizinische Hochschule Zentrum Frauenheilkunde Abt.Gynäkologische Onkologie, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Brustzentrum Rhein-Ruhr Servicegesellschaft mbH, Mönchengladbach
  - St. Vincenz-Krankenhaus GmbH Paderborn Frauen- und Kinderklinik St. Louise, Paderborn
- Italy (4):
  - A.O. S. Anna e San Sebastiano, Caserta, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Ospedale San Raffaele, Milan, Lombardy
  - Ospedale Santa Chiara, Trento, Trentino-Alto Adige
- Mexico (9):
  - Panamerican Clinical Research S.A de C.V., Guadalajara, Jalisco
  - RENATI INNOVATION S.A.P.I. de C.V, Guadalajara, Jalisco
  - COI Centro Oncologico Internacional Santa Fe, Mexico City, Mexico CITY (federal District)
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - OncoMed, Mexico City, Mexico CITY (federal District)
  - ARKE Estudios Clínicos S.A. de C.V., Mexico City, Mexico CITY (federal District)
  - Instituto Nacional de Cancerologia, Distrito Federal
  - CENEIT Oncologicos, Mexico City
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Morelia
- Poland (7):
  - Centrum Onkologii im. Prof. Franciszka ?ukaszczyka, Bydgoszcz
  - Narodowy Instytut Onkologii Odzia? w Gliwicach, Gliwice
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Szpital Wojewódzki im. Miko?aja Kopernika, Koszalin
  - Szpital Uniwersytecki w Krakowie, Krakow
  - MRUKMED Lekarz Beata Madej-Mruk i Partner Spolka Partnerska Oddzial nr 1 w Rzeszowie, Rzeszów
  - Narodowy Instytut Onkologii im. M.Sklodowskiej-Curie, Warsaw
- South Africa (2):
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Richards Bay Oncology Centre, KwaZulu Natal
- South Korea (10):
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (8):
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital San Pedro De Alcantara, Cáceres
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (6):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hosipital at Linkou, Taoyuan
  - Veterans General Hospital - Taichung, Xitun Dist.
  - National Taiwan University Hospital, Zhongzheng Dist.
- Turkey (Türkiye) (10):
  - Gulhane Training and Applicaton Hospital, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Dicle University Faculty of Medicine, Diyarbakır
  - Trakya University Medical Faculty, Edirne
  - Medipol Mega Üniversite Hastanesi Göztepe, Istanbul
  - Marmara Uni Faculty of Medicine, Istanbul
  - Ege Uni Medical Faculty Hospital, Izmir
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Goztepe Prof.Dr. Suleyman Yalcin City Hospital, Kadiköy
  - Hacettepe Uni Medical Faculty Hospital, Sihhiye/Ankara
- United Kingdom (9):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Blackpool Victoria Hospital, Blackpool
  - Western General Hospital, Edinburgh
  - Princess Alexandra Hospital, Harlow
  - St Bartholomew's Hospital, London
  - Maidstone & Tonbridge Wells Hospital, Maidstone
  - Mount Vernon & Watford Hospital Trust, Northwood
  - Churchill Hospital, Oxford
  - Royal Hampshire County Hospital, Winchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing